CLINICAL TRIAL: NCT06628921
Title: The Effectiveness of Eptinezumab During a Migraine Attack (the BE-FREE Study)
Acronym: BEFREE
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Società Italiana per lo Studio delle Cefalee (Other); Fondazione Policlinico Universitario Campus Bio-Medico (Other); SISC RICe Group (Unknown)
Responsible Party: Principal Investigator, Luigi Francesco Iannone, Researcher, University of Florence
Other Study IDs: Rice_5.1
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: headache; Pain; migraine; Eptinezumab
MeSH Terms: conditions — Migraine Disorders; Headache; Pain | interventions — eptinezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Episodic migraine: Patients affected by migraine with an episodic pattern (< 15 monthly migraine days) with or without aura according to ICHD-III criteria with ongoing migraine attack.
  Interventions: Drug: Eptinezumab 100 or 300 mg ev
- Chronic migraine: Group/Cohort Description: atients affected by chronic migraine (> 15 monthly headache days with at least 8 days with migraine features) according to ICHD-III criteria with ongoing migraine attack.
  Interventions: Drug: Eptinezumab 100 or 300 mg ev

INTERVENTIONS:
Drug: Eptinezumab 100 or 300 mg ev — Eptinezumab administered for migraine prevention in patients but with ongoing migraine attacks.
  Other Names: Eptinezumab

SUMMARY:
A perspective and multicentric study to evaluate the efficacy of eptinezumab administered during a migraine attack. During the intravenous infusion of eptinezumab, some patients experiencing an ongoing migraine attack report its resolution. This finding is known in the literature, having been described in the RELIEF study. This study was designed to also evaluate, in a real-world setting, the efficacy of eptinezumab in resolving the ongoing attack and the time frame within which the attack is resolved.

The study includes all patients who will begin treatment according to clinical practice, and are included in the TACHIS study (NCT06409845, Unique protocol ID RICe_5)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the third edition of the ICHD (ICHD-III).
* At least 8 days of migraine per month.
* Adequate compliance with study procedures.
* Availability of a migraine diary for at least one month prior to enrollment.
* Ongoing attack before administration.
* Included in the TACHIS study (NCT06409845)

Exclusion Criteria:

* Subjects with contraindications to the use of eptinezumab.
* Concomitant diagnosis of medical conditions and/or comorbidities that, in the investigator's opinion, could interfere with the study's assessments and outcomes.
* Pregnancy and breastfeeding.
* Changes in concomitant preventive therapy in the month prior to the initiation of eptinezumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multicentric study on patients attending the outpatient clinic of Italian Headache centres who meet criteria for eptinezumab use as migraine preventive treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Time to Headache Pain Freedom | Up to 48 hours postdose
  Time to headache pain freedom defined as the time that the participant reported freedom of pain, meaning their headache pain had gone from moderate to severe at baseline to no pain.

SECONDARY OUTCOMES:
Time to Absence of Most Bothersome Symptom (MBS) | Up to 48 hours postdose
  Time to absence of most bothersome symptom defined as the time that the participant reported absence of MBS
Headache Pain Freedom at 2 Hours | 2 hours
  Number of participants with freedom from headache pain at 2 hours postdose are reported.
Absence of MBS at 2 Hours | 2 hours
  Number of participants with absence of MBS (of nausea, photophobia, or phonophobia) at 2 hours postdose are reported.
Headache Pain Freedom and absence of MBS | Up to 48 hours postdose
  Number of participants with freedom from headache pain and/or Number of participants with absence of MBS up to 48 hours
Use of Rescue Medication | Up to 48 hours postdose
  Number of participants who used rescue medication up to 48 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Biomedico, Roma, Italy

REFERENCES:
- [Background] Winner PK, McAllister P, Chakhava G, Ailani J, Ettrup A, Krog Josiassen M, Lindsten A, Mehta L, Cady R. Effects of Intravenous Eptinezumab vs Placebo on Headache Pain and Most Bothersome Symptom When Initiated During a Migraine Attack: A Randomized Clinical Trial. JAMA. 2021 Jun 15;325(23):2348-2356. doi: 10.1001/jama.2021.7665. PMID 34128999